CLINICAL TRIAL: NCT02591680
Title: The Effect of Muscle Strengthening Associated With Neuromuscular Stimulus in Patients With Patellofemoral Pain During Negotiating Stairs: A Randomized Controlled Trial
Brief Title: The Effect of Muscle Strengthening Associated With Neuromuscular Stimulus in Patients With Patellofemoral Pain During Negotiating Stairs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Paulo Roberto Garcia Lucareli, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL004
Record Dates: First submitted 2015-10-26; First posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuromuscular training (Experimental): Neuromuscular, this arm will receive neuromuscular training and muscle strengthening.
  Interventions: Other: Neuromuscular training; Device: Sensorimotor
- Strength (Active Comparator): Strength, this arm will receive only muscle strengthening.
  Interventions: Other: Muscle strengthening

INTERVENTIONS:
Other: Neuromuscular training
  Other Names: Sensorimotor, balancing exercises, proprioceptive stimuli.
  Arms: Neuromuscular training
Other: Muscle strengthening
  Other Names: Hip abductors and lateral rotators and knee extensors strengthening
  Arms: Strength
Device: Sensorimotor
  Arms: Neuromuscular training

SUMMARY:
Assess pain, function, hip and knee strength and kinematics of trunk and lower limbs during ascent and descent stairs after the addition of neuromuscular training to hip muscle strengthening.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women,
* previous knee pain last 3 months in at least two of the following activities: sitting for long periods, walk up or down stairs, squat, running and jumping

Exclusion Criteria:

* Lower limb surgery,
* patella displacement
* knee instability
* Heart or locomotor disorders which might influence the evaluation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
3D kinematic range of motion of hip adduction during ascending and descending stairs | 4 weeks
  Kinematic analysis during ascent and descent stairs
3D kinematic range of motion of hip internal rotation during ascending and descending stairs | 4 weeks
  Kinematic analysis during ascent and descent stairs

SECONDARY OUTCOMES:
Pain Scores on the Numerical Pain Rating Scale | 4 weeks
Strength of hip and knee extensor muscles measured through hand-held dynamometer | 4 weeks
Lower Limb Function measured through the questionnaires Anterior Knee Pain Scale -AKPS and Functional Index Questionnaire- FIQ . | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Nove de Julho, São Paulo, São Paulo, Brazil